CLINICAL TRIAL: NCT00804843
Title: A Randomized Clinical Trial to Evaluate the Effects of High Dose Statin and Niacin Therapy on Excised Plaque Biomarkers in Patients Undergoing Carotid Endarterectomy (CEA)
Brief Title: Merck Carotid Atherosclerosis Trial (MK-0000-111)(COMPLETED)
Acronym: MCAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-111; 2008_598 (Other: Merck Study Number)
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Atorvastatin; Niacin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statin 80 mg + Niacin extended-release (ER) (Experimental): Participants in Russia and Brasil will receive 80 mg Simvastatin + niacin. All other participants will receive 80 mg Atorvastatin + niacin.
  Interventions: Drug: Atorvastatin/niacin extended-release; Drug: Simvastatin
- Statin 10 mg (Active Comparator): Participants in Russia and Brasil will receive 10 mg Simvastatin. All other participants will receive 10 mg Atorvastatin.
  Interventions: Drug: Atorvastatin; Drug: Simvastatin

INTERVENTIONS:
Drug: Atorvastatin/niacin extended-release — 80 mg tablet atorvastatin once daily, 10 mg tablet placebo to atorvastatin once daily, and niacin extended-release tablet starting at 500 mg daily and titrating to 2g daily. Treatment will be from 4 to 12 weeks.
  Other Names: Lipitor, Niaspan
  Arms: Statin 80 mg + Niacin extended-release (ER)
Drug: Atorvastatin — 10 mg tablet atorvastatin once daily, 80 mg tablet placebo to atorvastatin once daily, and placebo to niacin extended-release tablet starting at 500 mg daily and titrating to 2g daily. Treatment will be from 4 to 12 weeks.
  Other Names: Lipitor
  Arms: Statin 10 mg
Drug: Simvastatin — (Russia and Brazil) 80 mg tablet simvastatin once daily, 10 mg tablet placebo to simvastatin once daily, and niacin extended-release tablet starting at 500 mg daily and titrating to 2g daily. Treatment will be from 4 to 12 weeks.
  Other Names: Zocor
  Arms: Statin 80 mg + Niacin extended-release (ER)
Drug: Simvastatin — (Russia and Brazil) 10 mg tablet simvastatin once daily, 80 mg tablet placebo to simvastatin once daily, and placebo to niacin extended-release tablet starting at 500 mg daily and titrating to 2g daily. Treatment will be from 4 to 12 weeks.
  Other Names: Zocor
  Arms: Statin 10 mg

SUMMARY:
This study will examine the effect of statin and niacin therapy on carotid plaque biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with carotid stenosis AND is scheduled to undergo carotid endarterectomy
* Female patients of reproductive potential must abstain from sex or use an acceptable method of birth control through out the study

Exclusion Criteria:

* Patient must undergo CEA less than 4 weeks after entering study
* Patient has recent history of acute coronary syndrome
* Patient has has coronary artery bypass graft surgery within 30 days of study start
* Patient has thyroid disease that has not been treated for more than 6 weeks
* Patient has donated blood within 8 weeks of study start
* Patient has poorly controlled diabetes mellitis
* Patient has human immunodeficiency virus (HIV) or Hepatitis B or C
* Patient is taking warfarin or other anticoagulants
* Patient is taking hormone replacement therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Statin 80 mg + Niacin Extended-release (ER) | Statin 10 mg
Started | 50 | 50
Completed | 40 | 43
Not Completed | 10 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 8 | 5
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Statin 80 mg + Niacin ER: Participants in Russia and Brasil will receive 80 mg Simvastatin + niacin. All other participants will receive 80 mg Atorvastatin + niacin.
- Total: Total of all reporting groups
Arm/Group | Statin 80 mg + Niacin ER | Statin 10 mg | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.68 (9.42) | 69.20 (8.63) | 69.47 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 35 | 33 | 68

OUTCOME MEASURES:

1. Primary Outcome: Composite Score of Plaque Inflammation/Stability Gene Expression as Assayed by Ribonucleic Acid (RNA) Taqman Analysis
Description: Excised carotid plaques were evaluated for the gene expression of 60 biomarkers associated with inflammation ("Hot" biomarkers) & 25 biomarkers associated with stability ("Cold" biomarkers). Each biomarker was assayed using a quantitative polymerase chain reaction method and results were reported as a Cycle Threshold, (Ct). A Composite Score was calculated by averaging the Ct for each of the 25 "cold" genes, and subtracting the average Ct for the 60 "hot" genes. A higher composite score was associated with greater inflammation and a lower score was associated with stability (non-inflamed).
Time Frame: At time of carotid endarterectomy (after 4 to 12 weeks of dosing)
Population: Only participants who completed the study, had evaluable plaque samples and were at least 80% compliant with dosing schedule were included in the analysis.
Measure: Mean (Standard Deviation); unit: Cycle threshold (Ct)
Arm/Group | Statin 80 mg + Niacin Extended-release (ER) | Statin 10 mg
Number analyzed (Participants) | 36 | 34
Cycle threshold (Ct) | 1.36 (1.17) | 0.82 (1.33)
Statistical Analysis 1: Comparison: Statin 80 mg + Niacin Extended-release (ER) vs Statin 10 mg; Test type: Superiority or Other; p = 0.811, ANOVA; Least Square Mean Difference = 0.27, 90% CI 2-sided [-0.24 to 0.78]

2. Primary Outcome: Plaque Instability Protein Composite Score
Description: Each excised plaque was analyzed using an assay of 20 proteins that reflect plaque composition and inflammation. Each protein was assigned scaled signs, with a lower (negative) sign associated with plaque stability and a higher (positive) sign associated with plaque inflammation/instability. The Composite Score was the average amounts of all the 20 proteins with their associated signs. A higher Composite Score is associated with more plaque instability.
Time Frame: At time of carotid endarterectomy (after 4 to 12 weeks of dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Statin 80 mg + Niacin Extended-release (ER) | Statin 10 mg
Number analyzed (Participants) | 36 | 34
Score | -7.19 (10.45) | -10.48 (11.70)
Statistical Analysis 1: Comparison: Statin 80 mg + Niacin Extended-release (ER) vs Statin 10 mg; Test type: Superiority or Other; p = 0.898, ANOVA; Least Square Mean Difference = 3.64, 90% CI 2-sided [-1.09 to 8.36]

3. Primary Outcome: Total Cholesterol and Free Cholesterol Measured by Enzymatic Chromogenic Assay
Description: Cholesterol ester was to be calculated by the following formula: Cholesterol Ester = Total Cholesterol - Free Cholesterol.
Time Frame: At time of carotid endarterectomy (after 4 to 12 weeks of dosing)
Population: Only participants who completed the study, had evaluable plaque samples and were at least 80% compliant with dosing schedule were to be included in the analysis. This was not performed due to technical concerns. Instead, the cholesterol content determination, if performed, will use mass spectrometry approach and would be an exploratory objective.
Arm/Group | Statin 80 mg + Niacin Extended-release (ER) | Statin 10 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Statin 80 mg + Niacin Extended-release (ER): Participants in Russia and Brasil will receive 80 mg Simvastatin + niacin. All other participants will recieve 80 mg Atorvastatin + niacin
- Statin 10 mg: Participants in Russia and Brasil will receive 10 mg Simvastatin. All other participants will
  recieve 10 mg Atorvastatin.
Arm/Group | Statin 80 mg + Niacin Extended-release (ER) | Statin 10 mg
Serious Adverse Events (participants affected / at risk) | 9/50 | 7/50
Other Adverse Events (participants affected / at risk) | 5/50 | 2/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Statin 80 mg + Niacin Extended-release (ER) (N=50) | Statin 10 mg (N=50)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Chronic (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Statin 80 mg + Niacin Extended-release (ER) (N=50) | Statin 10 mg (N=50)
Flushing (Vascular disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications derived from the study should include input from the investigator(s) and SPONSOR. After to the multicenter publication, or 24 months after completion of the study, whichever comes first, an investigator may publish the results for the study site independently. The SPONSOR must have the opportunity to review all proposed publications 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.